CLINICAL TRIAL: NCT01809418
Title: Efficacy Study of the keePAP Device in Reducing the Number of Obstructive Breathing Events
Brief Title: keePAP Device for Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: keepMED Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: keePAP-1.0
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- keePAP (Experimental)
  Interventions: Device: keePAP

INTERVENTIONS:
Device: keePAP

SUMMARY:
The aim of the study is to test the hypothesis that a new device would produce a significant decrease in obstructive breathing events during sleep as indexed by the Apnea Hyperpnoea Index (AHI) or Respiratory Disturbance Index (RDI) and measures of oxygen saturation during sleep.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) syndrome is a disorder characterized by repetitive episodes of upper airway obstruction that occur during sleep. Associated features include loud snoring and fragmented non-refreshing sleep and have profound impact on quality of life, on safety on the roads and at work, and on the cardiovascular and metabolic systems.

The aim of the study is to test the hypothesis that a new device would produce a significant decrease in obstructive breathing events during sleep as indexed by the AHI/RDI and measures of oxygen saturation during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age over between 18 and 80 years old;
* AHI/RDI > 5

Exclusion Criteria:

* Uncontrolled or serious illness (angina/myocardial infarction, cancer, stroke, dementia, congestive heart failure),
* Exhibiting any flu-like or upper respiratory illness symptoms at time of assessment;
* History of severe nasal allergies or sinusitis or difficulty breathing through the nose;
* Persistent blockage of one or both nostrils;
* Any previous operation or trauma to the nose;
* Any nasal, facial or head abnormalities that would not allow adequate placement of the device.
* Previous diagnosis of insomnia, narcolepsy, periodic limb movement disorder, respiratory failure.
* Female subjects of childbearing age were excluded if they were pregnant or intending to become pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
AHI/RDI and oxygen saturation during sleep | one night
  Efficacy of the keePAP system in reducing the number of obstructive breathing events during sleep as indexed by the AHI and measures of oxygen saturation during sleep.

SECONDARY OUTCOMES:
Patient comfort | one night
  Patients will be asked to report their sleep experience and if any difficulties or discomfort was encountered.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601